CLINICAL TRIAL: NCT00903773
Title: A Phase I Open-label Trial to Investigate the Effect of Severe Renal Impairment on the Single-dose Pharmacokinetics of Telaprevir.
Brief Title: VX-950-TiDP24-C132: A Study to Investigate the Effect of Renal Impairment on the Pharmacokinetics of Telaprevir.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tibotec BVBA (Industry)
Responsible Party: Senior Director Compound Development Team Leader, Tibotec Pharmaceuticals, Ireland
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR016123
Record Dates: First submitted 2009-05-14; First posted 2009-05-18 (Estimated); Last update posted 2010-12-17 (Estimated); Status verified 2010-12

CONDITIONS: Hepatitis C; Kidney Diseases
Keywords: VX-950-TiDP24-C132; VX-950-C132; VX-950; HCV
MeSH Terms: conditions — Hepatitis C; Kidney Diseases | interventions — telaprevir

INTERVENTIONS:
Drug: telaprevir

SUMMARY:
The purpose of this study is to investigate the effect of severe renal impairment or failure on the single-dose pharmacokinetics of telaprevir (TVR). Pharmacokinetics means how the drug is absorbed into the bloodstream, distributed in the body and eliminated from the body. In addition, the effect of severe renal impairment on the total and unbound plasma concentrations of the sum of TVR and its R-diastereomer VRT-127394 will be assessed. (Diastereomers are substances whose chemical structures are mirror images of each other). Finally, the short-term safety and tolerability of TVR in participants with severe kidney disease will be determined. The results of this study will guide dose recommendations for TVR in subjects with kidney disease.

DETAILED DESCRIPTION:
This is a Phase I, open-label trial to investigate the single-dose pharmacokinetics of telaprevir (TVR) in 12 participants with severe renal impairment (defined as creatinine clearance (CrCl) < 30 mL/min) as compared to 12 participants with normal renal function, matched for sex, race, age (± 10 years) and BMI (± 20%). Open-label means that the study doctor and the participants know what treatment will be assigned to them. All participants will receive a single 750-mg dose of TVR. Pharmacokinetic profiles of total TVR up to 24 hours postdose will be determined. A 24 hour urine collection test will be performed to estimate the CrCl. In addition, the effect of severe renal impairment on the total and unbound plasma concentrations of the sum of TVR and VRT-127394 will be assessed. Tolerability and safety of TVR will be assessed throughout the trial period. Illnesses and side effects will be checked at every visit. Blood and urine samples will be taken at screening, on Day 1, 2 and at the 2 follow-up visits. ECG and vital signs will be taken at screening, twice on day 1, on day 2 and at the first follow-up visit. At the second follow-up visit vital signs alone will be determined. A physical examination will be done at screening, on the day before TVR intake, on day 2 and at both follow-up visits. All participants will receive a single 750-mg dose of telaprevir (TVR) given by mouth as 2 tablets of 375 mg.

ELIGIBILITY:
Inclusion Criteria:

* Males are allowed and females of childbearing potential if adequate contraception is used. Females of non-childbearing potential should be amenorrheal for at least 2 years, or have undergone tubal ligation (or other permanent birth control methods), or hysterectomy (total), or oophorectomy (bilateral)
* For participants with severe renal impairment: consistent with the disease process of chronic renal failure and associated symptoms, otherwise judged to be in good health in the opinion of the investigator on the basis of a medical evaluation (including a physical examination, medical history, electrocardiogram (ECG), vital signs, and screening laboratory tests), with any concomitant medical conditions under stable medical control
* For participants with severe renal impairment: creatinine clearance < 30 mL/min (Cockcroft-Gault)
* For healthy controls: healthy on the basis of a medical evaluation that reveals the absence of any clinically relevant abnormality and includes a physical examination, medical history, ECG, vital signs, and the results of blood biochemistry, blood coagulation and hematology tests and a urinalysis carried out at screening

Exclusion Criteria:

* A history of any illness (unrelated to renal impairment, as appropriate) that, in the opinion of the investigator, might confound the results of the study or pose an additional risk in administering study medication to the participant. This may include but is not limited to: diabetes mellitus, history of relevant drug or food allergies
* history of cardiovascular or central nervous system disease
* history or presence of clinically significant pathology, chronic skin disease, or history of mental disease
* For subjects with severe renal impairment: history of renal transplant or renal carcinoma. Participants with a history of renal carcinoma who have been cancer free for at least 5 years may be included
* For participants with severe renal impairment: participants with End Stage Renal Disease (ESRD) requiring dialysis
* For healthy controls: current use of prescription medication and regular treatment with over-the-counter medications

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2009-06; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
The primary objective of this study is to investigate the effect of severe renal impairment on the single-dose pharmacokinetics of total telaprevir. Total telaprevir is the sum of telaprevir bound to plasma proteins and unbound (free) telaprevir. | Pharmacokinetic profiles of total TVR up to 24 hours postdose will be determined. Twenty-four hour urine will be collected for estimation of CrCl.

SECONDARY OUTCOMES:
The effect of severe renal impairment on total and unbound plasma concentrations of the sum of TVR and VRT-127394 will be investigated. | Blood samples will be taken at specific timepoints within the 24-hour postdose period.
Safety and tolerability of a single dose of telaprevir will be determined. | This will be determined throughout the study.

CONTACTS AND LOCATIONS:
Overall Officials: Tibotec-Virco Virology BVBA Clinical Trial, Study Director — Tibotec BVBA